CLINICAL TRIAL: NCT04585607
Title: Long-term Effects of Expanded Hemodialysis in Reduction of Large Middle Molecules in Chronic Hemodialysis Patients: Potential Benefits to the Prevention of Sarcopenia
Brief Title: Potential Benefits of Expanded Hemodialysis in Prevention of Sarcopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hyeongcheon Park, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2020-0337
Record Dates: First submitted 2020-09-28; First posted 2020-10-14 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis

STUDY DESIGN:
Intervention Model Description: The participant hospital currently has around 90 maintenance HD patients and it is possible to recruit 74 patients for this study. Study subjects will be randomized to each treatment arm using a random number table. As outlined in the proposal, it is estimated that we may experience up to 30% of drop out during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expanded hemodialysis (HDx) (Experimental): HDx therapies be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription
  Interventions: Device: A medium cut-off dialyzer (Theranova) will be used for HDx.
- Conventional hemodialysis (Active Comparator): Conventional hemodialysis therapies be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription
  Interventions: Device: A synthetic high-flux dialyzer (Polyflux)

INTERVENTIONS:
Device: A medium cut-off dialyzer (Theranova) will be used for HDx. — A medium cut-off dialyzer used for HDx (Theranova) must be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required. General rules will be applied regarding dialysis prescription.
  HD with MCO dialyzer (Theranova 400®, Baxter) vs. high-flux dialyzer (eg. Polyflux H, Baxter)
  Arms: Expanded hemodialysis (HDx)
Device: A synthetic high-flux dialyzer (Polyflux) — A synthetic high-flux dialyzer (Polyflux) used for hemodialysis must be implemented following current clinical practices guidelines and procedures at the hospital. No additional actions are required.
  Arms: Conventional hemodialysis

SUMMARY:
The current study will investigate whether long term implementation of expanded hemodialysis (HDx) will effectively decrease serum levels of large uremic toxins and ameliorate progression of sarcopenia in patients with chronic kidney disease requiring hemodialysis.

DETAILED DESCRIPTION:
This is an open-label, prospective, 1:1 randomized, parallel-group, study to evaluate the efficacy of expanded hemodialysis (HDx) compared to conventional hemodialysis in patients with chronic kidney disease in South Korea for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* On HD treatment over 6 months before study enrollment
* Aged over 18 years
* Able to give informed consent

Exclusion Criteria:

1. Hemiplegia or paraplegia state
2. Planned renal transplant or conversion to peritoneal dialysis within study period
3. Active chronic infection or inflammatory conditions including autoimmune disease, inflammatory arthritis and active malignancy
4. History of monoclonal gammopathy
5. Life expectancy <12 months
6. Pregnancy or breast feeding
7. Receiving immunosuppressant medication
8. Inability to complete study assessments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Biomarkers of sarcopenia | Changes in serum level of Myostatin and IGF-1 every 6 months
  Change in blood levels of myostatin and insulin-like growth factor-1 (IGF-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No